CLINICAL TRIAL: NCT01224236
Title: Randomized Trial Comparing Iron Supplementation Versus Routine Iron Intake in Very Low Birth Weight (VLBW) Infants
Brief Title: Randomized Trial of Iron Supplementation to Prevent Anemia in Very-low-birth-weight Infants
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Kathleen Kennedy, Professor - Pediatrics, Neonatology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCT of Iron Supplementation
Record Dates: First submitted 2010-10-14; First posted 2010-10-19 (Estimated); Results first posted 2015-06-19 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Iron-Dextran Complex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- iron supplementation (Experimental): 2 mg/kg/day of elemental iron as a multivitamin with iron solution
  Interventions: Drug: Iron Supplement
- control (Sham Comparator): multivitamin solution without iron
  Interventions: Drug: control

INTERVENTIONS:
Drug: Iron Supplement — 2 mg/kg/day elemental iron as multivitamin with iron solution
  Arms: iron supplementation
Drug: control — multivitamin solution without iron
  Arms: control

SUMMARY:
The purpose of this study is to determine if iron supplementation in addition to routine iron intake decreases the risk of developing anemia in preterm infants.

DETAILED DESCRIPTION:
Objective was to determine if iron supplementation of 2 mg/kg per day, in addition to routine iron-fortified formula or mother's milk, increased the hematocrit (Hct) at 36 weeks' postmenstrual age (PMA).

All infants have a decline in hemoglobin(Hgb) after birth because of increasing PaO2 and Hgb saturation after birth. In very low birth weight (VLBW) infants (birth weight ,1500 g), the nadir at 1 to 3 months after birth is lower than in term infants because of (1) greater phlebotomy losses for blood tests, (2) shortened red blood cell survival, and (3)rapid growth.

VLBW infants may be at increased risk of developing iron deficiency anemia because of (1) low iron stores at birth, (2) rapid depletion of iron stores owing to phlebotomy losses, and (3) inability to regulate iron absorption by the gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

1. birth weight: < 1500 grams
2. Tolerating iron fortified preterm formula or fortified breast milk at 120cc/kg/day by 8 weeks of age
3. ≤32 weeks adjusted post-menstrual age at the time of enrollment

Exclusion Criteria:

1. cyanotic heart disease
2. bowel resection prior to enrollment

Max Age: 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2010-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kennedy Kathleen, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Children's Memorial Hermann Hospital, Houston, Texas, United States

REFERENCES:
- [Result] Taylor TA, Kennedy KA. Randomized trial of iron supplementation versus routine iron intake in VLBW infants. Pediatrics. 2013 Feb;131(2):e433-8. doi: 10.1542/peds.2012-1822. Epub 2013 Jan 21. PMID 23339225

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants were screened by birth weight on admission to the neonatal intensive care unit (NICU). If birth weight criteria were met, infants were followed to see if they met eligibility criteria. If they approached eligibility, parents were approached for consent by the investigator. IRB approved to recruit 4/6/2010. Enrollment completed by 10/2012.
Pre-assignment Details: All groups started the study intervention once they had reached goal feedings of 120 cc/kg/day
Period: Overall Study
Arm/Group | Iron Supplementation | Control
Started | 76 | 74
Completed | 75 | 73
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iron Supplementation | Control | Total
Number analyzed (Participants) | 76 | 74 | 150
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Age is reported as postmenstrual age (PMA), which is the gestational age in weeks plus the postnatal age in weeks.
  weeks | 29.7 (1.5) | 29.7 (1.4) | 29.7 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 35 | 73
  Male | 38 | 39 | 77
Region of Enrollment [Number; unit: participants]
  United States | 76 | 74 | 150

OUTCOME MEASURES:

1. Primary Outcome: Hematocrit (Hct)
Description: For infants discharged from the hospital before 36 weeks' postmenstrual age (PMA), the last Hct before discharge was used. For infants transferred before 36 weeks PMA, the Hct at 36 weeks was sought from the receiving hospital and used if available. For infants transferred before 36 weeks with no available Hct at 36 weeks, the last Hct before transfer was used. For those who died before 36 weeks PMA, the Hct at 36 weeks was considered to be missing.
Time Frame: 36 weeks postmenstrual age (PMA)
Measure: Mean (Standard Deviation); unit: percentage of red blood cells in blood
Arm/Group | Iron Supplementation | Control
Number analyzed (Participants) | 75 | 73
percentage of red blood cells in blood | 29.2 (4) | 28.3 (4.5)

2. Secondary Outcome: Transfusions
Description: # of transfusions infants required after enrollment.
Time Frame: enrollment to 36 weeks postmenstrual age (PMA)
Measure: Median (Inter-Quartile Range); unit: transfusions
Arm/Group | Iron Supplementation | Control
Number analyzed (Participants) | 76 | 74
transfusions | 1 [0 to 2] | 1 [0 to 2]

ADVERSE EVENTS:
Arm/Group | Iron Supplementation | Control
Serious Adverse Events (participants affected / at risk) | 1/76 | 1/74
Other Adverse Events (participants affected / at risk) | 0/76 | 0/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron Supplementation (N=76) | Control (N=74)
death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) — Deaths are a possible and anticipated adverse event for this population. Neither death was related to study participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes